CLINICAL TRIAL: NCT06416995
Title: Investigation of First Trimester Serum Vasohibin-1, Vasohibin-2, Cardiotrophin-1 and Endocan Concentrations in Predicting Adverse Perinatal Outcomes
Brief Title: Serum Vasohibin, Cardiotrophin, Endocan & Perinatal Outcomes
Status: Recruiting | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ibrahim kale, Associate professor, Umraniye Education and Research Hospital
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01I 5q
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Preeclampsia; Gestational Hypertension; Gestational Diabetes; Preterm Birth; Fetal Growth Retardation
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Diabetes, Gestational; Premature Birth; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Pregnant women who do not have any pregestational disease, who gave a blood sample in the first trimester for the study, who did not develop any pregnancy-related disease during their pregnancy, and who gave birth at term.
  Interventions: Diagnostic Test: first trimester serum diagnostic test
- Adverse Perinatal Outcome Group: Pregnant women who do not have any pregestational disease and who gave a blood sample in the first trimester for the study and who develop preeclampsia, gestational hypertension, preterm birth, fetal growth restriction, and gestational diabetes mellitus in the later weeks of pregnancy.
  Interventions: Diagnostic Test: first trimester serum diagnostic test

INTERVENTIONS:
Diagnostic Test: first trimester serum diagnostic test — First trimester serum vasohibin-1, vasohibin-2, cardiotropin-1 and endocan concentrations predict adverse perinatal outcomes

SUMMARY:
Investigation of the relationship between maternal serum vasohibin-1, vasohibin-2, cardiotrophin -1 and endocan concentrations at the 11th and 14th weeks of gestation and adverse perinatal outcomes.

DETAILED DESCRIPTION:
Previous animal model studies in the literature have shown that vasohibin-1 released in endothelial cells inhibits angiogenesis, while vasohibin-2 stimulates angiogenesis. Additionally, immunohistochemical studies have shown that vasohibin-2 plays a role in the cellular fusion of trophoblasts in the placenta to form syncytiotrophoblasts.

Studies in the literature have shown that cardiotrophin-1 is expressed in cardiac myocytes and vascular endothelial cells and stimulates the synthesis and secretion of endothelin-1 in endothelial cells through the gp130 signaling pathway. Since endothelin 1 plays an important role in the regulation of vascular tone, cardiotrophin-1 can be considered to act as an endothelium-derived biological factor, possibly involved in the regulation of vascular tone under normal physiological conditions or secondary to pathological processes.

Studies in the literature have shown that maternal serum endocan levels are higher in pregnant women whose pregnancies were complicated by preeclampsia than in normotensive pregnant women, and that the endocan molecule may be effective in the etiopathogenesis of preeclampsia, especially if it develops early.

In the light of this above-mentioned information, we aim to investigate whether serum vasohibin-1, vasohibin-2, cardiotrophin-1 and endocan concentrations measured during the 11th to 14th weeks of pregnancy can be used to predict preeclampsia, gestational hypertension, fetal growth restriction, preterm birth and gestational diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Those who had the first-trimester screening test between 11 and 14 weeks of pregnancy and are in the low-risk group
* Those with singleton pregnancy
* Those who did not conceive pregnancy with assisted reproductive treatment methods
* Those who do not have any pregestational diseases
* Those who do not have any uterine anomalies

Exclusion Criteria:

* Smokers
* Those who are in the high-risk group with the first trimester screening test
* Those with multiple pregnancies
* Those who conceive with assisted reproductive treatment methods
* Those who had any disease before pregnancy
* Those who have any uterine anomalies

Ages: 18 Years to 39 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant women with a singleton pregnancy who are between 11 and 14 weeks of gestation, who do not smoke, and do not have any systemic disease.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Usability of serum vasohibin-1, vasohibin-2, cardiotropin-1 and endocan concentrations in predicting adverse perinatal outcomes | 1 year
  Usability of serum vasohibin-1, vasohibin-2, cardiotropin-1 and endocan concentrations in predicting adverse perinatal outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Ümraniye Eğitim ve Araştırma Hastanesi, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided